CLINICAL TRIAL: NCT06051214
Title: Thrombin Generation and Prediction of Thromboembolic Events in Oncology Patients At Risk
Acronym: THROMBIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: Diagnostica Stago (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICO-2022-19
Record Dates: First submitted 2023-08-31; First posted 2023-09-22 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Solid Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thrombogram (Experimental): Blood sampling every month for 12 months
  Interventions: Biological: thrombogram

INTERVENTIONS:
Biological: thrombogram — blood sampling every month for 12 months

SUMMARY:
Coagulation is a complex system which, through the action of thrombin, leads to the formation of fibrin, which stabilises the platelet clot. Any disturbance in the balance between procoagulant and anticoagulant factors can tip the physiological process either towards a state of hypercoagulability leading to thrombosis or hypocoagulability responsible for bleeding.

Due to a number of factors, cancer is associated with a state of hypercoagulability, leading to thrombosis. The incidence of venous thromboembolism (VTE) in cancer patients varies from 15 to 20% depending on the type of cancer, the stage of the disease and the associated treatments (ONCORIF data, November 2021). The risk of venous thromboembolism (VTE) is greatly increased in cancer patients (RR x 3 to 6) and doubled in the case of associated chemotherapy (1). VTE is a poor prognostic factor, occurs mainly in the first 6 months after diagnosis and is the second leading cause of death in cancer patients.

At present, haemostasis tests performed in medical laboratories independently explore the different coagulation pathways but do not allow the overall haemostatic profile of a hyper- or hypocoagulable patient to be assess.

Based on this knowledge base, the aim of our study will be to monitor thrombogram profiles during the management of patients with tumours at high risk of thromboembolism (lung, pancreas, stomach, glioblastoma) and to correlate these profiles with the risk of a thromboembolic event occurring in these patients. The aim of the project is to validate a simple predictive test (suitable for clinical use) for the risk of thromboembolism in these patients. These analyses will also make it possible to monitor the impact of chemotherapy on changes in the thrombin generation test in patients.

DETAILED DESCRIPTION:
Biological blood samples will be taken specifically for research purposes. As far as possible and depending on the patient's schedule, a sample will be taken every month (during a consultation and/or a course of chemotherapy) and for the 12 months following the initiation of systemic treatment

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged > 18 years,
2. Patient with a solid cancer at high risk of thrombosis, whether metastatic or not (lung, pancreatic, gastric or glioblastoma cancers)1,
3. Patients who have not received any systemic treatment for their cancer,
4. An informed patient who does not object to the use of data for research purposes and who has consented to the collection, use and storage of biological samples.

Exclusion Criteria:

1. Patient who has had a VTE in the 12 months preceding the diagnosis of cancer,
2. Patient on low molecular weight heparins, standard unfractionated heparins and anti-vitamin K2,
3. Women who are pregnant, likely to become pregnant or who are breast-feeding,
4. Persons deprived of their liberty, under court protection, under curators or under the authority of a guardian,
5. Unable to undergo medical monitoring of the trial for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
To assess whether changes in thrombogram values are predictive of thromboembolic events in patients with solid cancers in the 12 months following initiation of their systemic treatment. | 12 months
  Venous thromboembolism (VTE)-free survival.

SECONDARY OUTCOMES:
Describe kinetic evolution of thrombogram after different chemotherapies | Every 3 months for 12 months
  Area Under the Curve/ Endogenous Thrombin Potential(ETP) (nM.min)
Describe kinetic evolution of thrombogram in metastatic disease | Every 3 months for 12 months
  Analysis of Area Under the Curve/ Endogenous Thrombin Potential(ETP) (nM.min) will be done before and after metastatic progression, or at each progression for patients with immediate metastatic disease.
Identify specific patterns of thrombogram evolution over time | Every 3 months for 12 months
  Homogeneous patient trajectories will be identified by evolution of Area Under the Curve/ Endogenous Thrombin Potential(ETP) (nM.min)

CONTACTS AND LOCATIONS:
Overall Officials: Judith RAIMBOURG, MD, Principal Investigator — INSTITUT DE CANCEROLOGIE DE L'OUEST
Locations (1):
- Institut de Cancerologie de L'Ouest, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No